CLINICAL TRIAL: NCT05851170
Title: Use of Warm Compresses During the Second Stage and the Risk of Perineal Tears: a Randomized Controlled Trial
Brief Title: Use of Warm Compresses During the Second Stage and the Risk of Perineal Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr Raneen Abu Shqara, Principal investigator, clinical instructor, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHR-0198-22
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Perineum; Tear
Keywords: Perineal tear; Warm compresses; Intact perineum; Almond oil
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of warm compresses and almond oil use during the second stage (Experimental): Warm compresses will be attached to the perineum between pushing During active pushing - almond oil will be used on the perineum (our routine care).
  Interventions: Other: The use of warm compresses and almond oil on the perineum during second stage
- Use of almond oil use (routine care) during the second stage (Active Comparator): During active pushing - almond oil will be applied on the perineum
  Interventions: Other: Use of almond oil use (routine care) during second stage

INTERVENTIONS:
Other: The use of warm compresses and almond oil on the perineum during second stage — Hot water from the tap at a temperature of (45-590c) will be poured into a container, and will be changed every 15 minutes.
  Timing of the start: when the baby's head descends in the pelvic canal and the woman feels the need to push The intervention: warm compresses will be attached to the perineum between the pressures During the pressing - almond oil will be applied. Meanwhile, the compresses will be returned to a bowl containing hot water. Every 15 minutes until birth the water will be replaced with hot water at an initial temperature of 45-590c.
  It is necessary to use compresses for a minimum of 10 minutes, and a maximum of 30 minutes.
  Other Names: Experimental
  Arms: Use of warm compresses and almond oil use during the second stage
Other: Use of almond oil use (routine care) during second stage — Routine care in the department is the use of almond oil during the second stage of pregnancy, during pushing.
  Other Names: Routine care
  Arms: Use of almond oil use (routine care) during the second stage

SUMMARY:
There is a controversy regarding whether warm compresses influence the rate of intact perineum after a vaginal delivery.

According to a meta-analysis published in 2019 that included 7 randomized prospective trials, approximately 2103 participants, the use of warm compresses during the second stage of labor increased the chance of an intact perineum RR=1.46, decreased the chance of a third degree tear RR=0.38 and grade four tear RR=0.11. The limitations noted in this meta-analysis include non-uniformity in the methods of the studies included in the meta-analysis in terms of the number of participants, the duration of use of the compresses, and the temperature of the compresses. In summary, it is reported that there is a need for more randomized studies.

Since there is a need for more randomized studies in the field, the study's goal is to conduct a randomized study that will compare the use of warm compresses in the second stage of labor against a standard care control group (almond oil) - in terms of perineal tear that will require suturing.

DETAILED DESCRIPTION:
Various techniques have been developed to prevent the development of perineal tears. As reported in the literature, active protection of the perineum during the second stage of labor can reduce the rate of tears. These include massage of the perineum, hands-on technique, use of gel, and warm compresses.

According to a Cochrane review that examined the use of warm compresses published in 2017, there is no difference in terms of the rate of events of an intact perineum, perineal trauma that requires suturing, but in a subanalysis it showed that there is a decrease in the rate of advanced tears, involving the anal sphincter and the rectal mucosa (grade three and four).

According to a meta-analysis published in 2019 that included 7 randomized prospective trials, approximately 2103 participants, the use of warm compresses during the second stage of labor increased the chance of an intact perineum RR=1.46, decreased the chance of a third degree tear RR=0.38 and grade four tear RR=0.11. The limitations noted in this meta-analysis include non-uniformity in the methods of the studies included in the meta-analysis in terms of the number of participants, the duration of use of the compresses, and the temperature of the compresses. In summary, it is reported that there is a need for more randomized studies.

Since there is a need for more randomized studies in the field, the study's goal is to conduct a randomized study that will compare the use of warm compresses in the second stage of labor against a standard care control group (almond oil) - in terms of perineal tear that will require suturing.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Singleton pregnancy
* Vertex presentation

Exclusion Criteria:

* Women with a history of third degree perineal tear in the past
* Intrauterine fetal death
* Crohn disease with perineal involvement

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 412 (Estimated)
Dates: Start 2023-06-11 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with perineal tear | 2 years
  Perineal tear (spontaneous) that required suturing

SECONDARY OUTCOMES:
Number of patients with episiotomy | 2 years
  The rate of episiotomy
Number of patients with mild perineal tear | 2 years
  First and second degree
Number of patients with with advanced perineal tear | 2 years
  Third and fourth degree

CONTACTS AND LOCATIONS:
Overall Officials: Raneen Abu Shqara, MD, Principal Investigator — Galilee Medical Center
Locations (1):
- Galilee Medical Center, Nahariya, Northern District, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aasheim V, Nilsen ABV, Reinar LM, Lukasse M. Perineal techniques during the second stage of labour for reducing perineal trauma. Cochrane Database Syst Rev. 2017 Jun 13;6(6):CD006672. doi: 10.1002/14651858.CD006672.pub3. PMID 28608597
- [Background] Magoga G, Saccone G, Al-Kouatly HB, Dahlen G H, Thornton C, Akbarzadeh M, Ozcan T, Berghella V. Warm perineal compresses during the second stage of labor for reducing perineal trauma: A meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2019 Sep;240:93-98. doi: 10.1016/j.ejogrb.2019.06.011. Epub 2019 Jun 15. PMID 31238205
- [Background] Pierce-Williams RAM, Saccone G, Berghella V. Hands-on versus hands-off techniques for the prevention of perineal trauma during vaginal delivery: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2021 Mar;34(6):993-1001. doi: 10.1080/14767058.2019.1619686. Epub 2019 Jun 3. PMID 31092083
- [Background] Geranmayeh M, Rezaei Habibabadi Z, Fallahkish B, Farahani MA, Khakbazan Z, Mehran A. Reducing perineal trauma through perineal massage with vaseline in second stage of labor. Arch Gynecol Obstet. 2012 Jan;285(1):77-81. doi: 10.1007/s00404-011-1919-5. Epub 2011 May 26. PMID 21614497